CLINICAL TRIAL: NCT01191255
Title: A Three-Period, 58-Week Safety and Efficacy Trial of KRX-0502 (Ferric Citrate) in Patients With End-Stage Renal Disease (ESRD) on Dialysis
Brief Title: A 58-Week Safety and Efficacy Trial of Ferric Citrate in Patients With ESRD on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KRX-0502-304; NCT01510106 (obsolete NCT alias)
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Hyperphosphatemia; Kidney Failure
Keywords: ESRD; end-stage renal disease; dialysis; hemodialysis; peritoneal dialysis; hemodialysis (HD); peritoneal dialysis (PD); chronic renal insufficiency; phosphate binder; kidney failure; renal failure
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — ferric citrate; Sevelamer; calcium acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Control (Active Comparator): PhosLo (calcium acetate) Renvela (sevelamer carbonate)
  Interventions: Drug: ferric citrate, ca acetate, sevelamer carbonate, placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: ferric citrate, ca acetate, sevelamer carbonate, placebo
- KRX-0502 (Ferric Citrate) (Experimental): ferric citrate
  Interventions: Drug: ferric citrate, ca acetate, sevelamer carbonate, placebo

INTERVENTIONS:
Drug: ferric citrate, ca acetate, sevelamer carbonate, placebo — All intervention doses will be based on serum phosphorus levels and/or drug label requirements
  Other Names: PhosLo; Renvela; KRX-0502; Zerenex

SUMMARY:
This is up to a 58 week study comparing ferric citrate to active control for 52 weeks in ESRD dialysis patients, and subsequently comparing ferric citrate to placebo for 4 weeks.

DETAILED DESCRIPTION:
This trial is a three-period, multicenter, safety and efficacy clinical trial. The first period is a two-week Washout Period, the second period is a 52-week randomized, open-label, active control Safety Assessment Period, and the third period is a four-week, randomized, open-label, placebo-controlled Efficacy Assessment Period in only the patients who were randomized to treatment with ferric citrate during the Safety Assessment Period. The primary objectives of this trial are to determine the long-term safety over 52 weeks of up to twelve (12) caplets/day of KRX-0502 (ferric citrate) in patients with ESRD undergoing either hemodialysis or peritoneal dialysis and to determine the efficacy of KRX-0502 (ferric citrate) in the four-week, randomized, open-label, placebo-controlled Efficacy Assessment Period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-breast-feeding females
2. Age ≥18 years
3. On thrice-weekly hemodialysis or on peritoneal dialysis for at least the previous three months prior to Screening
4. Serum phosphorus ≥6.0 mg/dL for study entry
5. Taking less than 3-18 pills/day of current phosphate binder
6. Willing to be discontinued from current phosphate binder(s) and initiated on ferric citrate
7. Willing and able to give informed consent
8. Life expectancy >1 year

Exclusion Criteria:

1. Parathyroidectomy within six months prior to Screening
2. Actively symptomatic gastrointestinal bleeding or inflammatory bowel disease
3. History of multiple drug allergies or intolerances
4. History of malignancy in the last five years (treated cervical or non-melanomatous skin cancer may be permitted if approved by CCC)
5. Previous intolerance to oral ferric citrate
6. Intolerance to oral iron-containing products
7. Psychiatric disorder that interferes with the patient's ability to comply with the study protocol
8. Inability to tolerate oral drug intake
9. Intolerance to calcium acetate and sevelamer carbonate
10. Any other medical condition that renders the patient unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the patient
11. Receipt of any investigational drug within 30 days of Screening Visit (Visit 0)
12. Inability to cooperate with study personnel or history of noncompliance
13. Unsuitable for this trial per Investigator's clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Lewis, MD, Study Chair — Collaborative Study Group; Samuel Blumenthal, MD, Study Chair — Collaborative Study Group
Locations (56):
- United States (52):
  - Southwest Clinical Research Institute, LLC, Tempe, Arizona
  - Tower Nephrology Medical Group, Los Angeles, California
  - Veterans Administration Greater Los Angeles Healthcare System, West Los Angeles, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - American Institute of Research, Whittier, California
  - University of Colorado Denver, Aurora, Colorado
  - Western Nephrology, Westminster, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Mayo Clinic, Jacksonville, Florida
  - ASA Clinical Research, LLC, Jupiter, Florida
  - Ocala Kidney Group, Ocala, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Atlanta Nephrology Referral Center, Decatur, Georgia
  - Circle Medical Management, Chicago, Illinois
  - Nephrology Specialists, PC, Michigan City, Indiana
  - LSU Health Sciences Center Section of Nephrology and Hypertension Department of Internal Medicine, New Orleans, Louisiana
  - Rockville Dialysis Center, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Pioneer Valley Nephrology, Holyoke, Massachusetts
  - Western New England Renal & Transplant Associates, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Kidney Consultants, PC, Pontiac, Michigan
  - Nephrology Hypertension Clinic, Southgate, Michigan
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Brookdale Physician's Dialysis Associates, Brooklyn, New York
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Duke University Medical Center Division of Nephrology, Durham, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Clinical Research Limited, Canton, Ohio
  - Division of Nephrology and Hypertension Department of Internal Medicine University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic Foundation Q7-150 Nephrology, Cleveland, Ohio
  - The Ohio State University Division of Nephrology, Columbus, Ohio
  - DaVita, Oklahoma City, Oklahoma
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Southeast Renal Research Institute Nephrology Associates, Chattanooga, Tennessee
  - Nephrology Associates, PC, Nashville, Tennessee
  - Vanderbilt University Medical Center Clinical Trials Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Kidney Associates, Houston, Texas
  - Nephrology, PA, Houston, Texas
  - Kidney Specialists of North Houston, PLLC, The Woodlands, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Vermont/ Fletcher Allen Health Care; Renal Services, Burlington, Vermont
  - Nephrology Clinical Research Center, Charlottesville, Virginia
  - Clinical Research & Consulting Center, LLC, Fairfax, Virginia
  - Nephrology Associates of Northern Virginia, Inc., Fairfax, Virginia
  - Peninsula Kidney Associates, Hampton, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Wisconsin Froedert Memorial Lutheran Hospital Division of Nephrology, Milwaukee, Wisconsin
- Israel (2):
  - Department of Nephrology and Hypertension Brazilai Medical Center, Ashkelon
  - Tel Aviv Sourasky Medical Center Nephrology Department, Tel Aviv
- Puerto Rico (2):
  - RCMI-Clinical Research Center Medical Sciences Campus University of Puerto Rico, Rio Piedras, PR
  - Puerto Rico Renal Health & Research Center, Inc/ Atlantic Healthcare Group, Inc, Trujillo Alto, PR

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Rodby RA, Umanath K, Niecestro R, Bond TC, Sika M, Lewis J, Dwyer JP; Collaborative Study Group. Ferric Citrate, an Iron-Based Phosphate Binder, Reduces Health Care Costs in Patients on Dialysis Based on Randomized Clinical Trial Data. Drugs R D. 2015 Sep;15(3):271-9. doi: 10.1007/s40268-015-0103-y. PMID 26239948
- See also: Sponsor Website — http://www.keryx.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Only subjects that completed the SAP on KRX-0502 were eligible to be included in the EAP
  2. in the EAP, subjects received only Placebo or KRX-0502-EAP
  3. 3 Subjects switched from 'Active Control' to KRX-0502 during the SAP and were randomized into the EAP
  4. In the 'Active Control' group, a combination of phosphate binders was allowed
Groups:
- Active Control-SAP: Patients received either PhosLo (calcium acetate), Renvela (sevelamer carbonate), or a combination of these treatments during a 52-week Safety Assessment Period.
- KRX-0502 (Ferric Citrate)-SAP: Patients received KRX-0502 (ferric citrate) during a 52-week Safety Assessment Period.
  Patients that completed the 52-week Safety Assessment Period were randomized to continue to receive KRX-0502 (ferric citrate) or placebo for a 4-week Efficacy Assessment Period.
- Placebo-EAP; KRX-0502 (Ferric Citrate)-EAP: Patients that completed the 52-week Safety Assessment Period on KRX-0502 were randomized 1:1 to continue to receive KRX-0502 (ferric citrate) or placebo for a 4-week Efficacy Assessment Period.
Period: Safety Assessment Period
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Started | 149 (3 subjects were assigned to receive KRX-0502 but didn't receive a single dose) | 292 | 0 | 0
Safety Population | 149 | 289 | 0 | 0
Completed | 111 | 193 | 0 | 0
Not Completed | 38 | 99 | 0 | 0
Period: Efficacy Assessment Period
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Started | 0 | 0 | 96 | 96
Completed | 0 | 0 | 70 | 90
Not Completed | 0 | 0 | 26 | 6

BASELINE CHARACTERISTICS:
Population: Total number of subjects in the full analysis population in the SAP was 427. 182 subjects that were treated with KRX-0502 in the SAP were randomized 1:1 to receive either KRX-0502 or Placebo in the EAP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP | Total
Number analyzed (Participants) | 146 | 281 | 91 | 91 | 609
Age, Customized [Number; unit: participants]
  Age <65 years (SAP) | 118 | 223 | 0 | 0 | 341
  Age >= 65 years (SAP) | 28 | 58 | 0 | 0 | 86
  Age <65 years (EAP) | 0 | 0 | 77 | 73 | 150
  Age >= 65 years (EAP) | 0 | 0 | 14 | 18 | 32
Sex/Gender, Customized [Number; unit: participants]
  Female (SAP) | 62 | 106 | 0 | 0 | 168
  Male (SAP) | 84 | 175 | 0 | 0 | 259
  Female (EAP) | 0 | 0 | 77 | 73 | 150
  Male (EAP) | 0 | 0 | 14 | 18 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino (SAP) | 23 | 41 | 0 | 0 | 64
  Not Hispanic or Latino (SAP) | 123 | 239 | 0 | 0 | 362
  Unknown or not reported (SAP) | 0 | 1 | 0 | 0 | 1
  Hispanic or Latino (EAP) | 0 | 0 | 14 | 9 | 23
  Not Hispanic or Latino (EAP) | 0 | 0 | 77 | 82 | 159
  Unknown or not reported (EAP) | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native (SAP) | 1 | 2 | 0 | 0 | 3
  Asian (SAP) | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander (SAP) | 2 | 0 | 0 | 0 | 2
  Black or African American (SAP) | 77 | 153 | 0 | 0 | 230
  White (SAP) | 61 | 114 | 0 | 0 | 175
  More Than One Race (SAP) | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported (SAP) | 4 | 11 | 0 | 0 | 15
  American Indian or Alaska Native (EAP) | 0 | 0 | 1 | 0 | 1
  Asian (EAP) | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander (EAP) | 0 | 0 | 0 | 0 | 0
  Black or African American (EAP) | 0 | 0 | 48 | 59 | 107
  White (EAP) | 0 | 0 | 39 | 28 | 67
  More Than One Race (EAP) | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported (EAP) | 0 | 0 | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Serum Phosphorus From Baseline (Week 52) to the End of the Efficacy Assessment Period (EAP; Week 56)
Description: Patients who completed the 52-week Safety Assessment Period (SAP) on KRX-0502 (ferric citrate) were randomized in a 1:1 ratio to receive either KRX-0502 (ferric citrate) or Placebo for 4 weeks.
Time Frame: 4 weeks
Population: Full Analysis Population (LOCF)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Number analyzed (Participants) | 0 | 0 | 91 | 91
mg/dL
  Baseline (Week 52) |  |  | 5.44 (1.459) | 5.12 (1.189)
  End of EAP (Week 56) |  |  | 7.23 (1.784) | 4.89 (1.291)
Statistical Analysis 1: Comparison: Placebo-EAP vs KRX-0502 (Ferric Citrate)-EAP; Test type: Superiority or Other; p < 0.0001, ANCOVA — The P-value for the change in mean serum phosphorus was calculated via an ANCOVA model with treatment as the fixed effect and Week-52-baseline as the co-variate

2. Secondary Outcome: Change in Mean Serum Ferritin From Baseline to Week 52
Time Frame: 52 weeks
Population: Full Analysis Population (LOCF)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Number analyzed (Participants) | 137 | 253 | 0 | 0
ng/mL
  Baseline | 609.50 (307.689) | 592.80 (292.863) |  |
  End of SAP (Week 52) | 631.87 (368.919) | 894.88 (481.788) |  |
Statistical Analysis 1: Comparison: Active Control-SAP vs KRX-0502 (Ferric Citrate)-SAP; Test type: Superiority or Other; p < 0.0001, ANCOVA — The P-value for the change in mean serum Ferritin were created via an ANCOVA model with treatment as the fixed effect and Study-baseline as the co-variate

3. Secondary Outcome: Change in Mean Serum Transferrin Saturation (TSAT) From Baseline to the End of the Safety Assessment Period (Week 52)
Time Frame: 52 weeks
Population: Full Analysis Population (LOCF)
Measure: Mean (Standard Deviation); unit: % Saturation
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Number analyzed (Participants) | 137 | 252 | 0 | 0
% Saturation
  Baseline | 30.8 (11.57) | 31.3 (11.21) |  |
  End of SAP (Week 52) | 29.7 (11.43) | 39.2 (16.78) |  |
Statistical Analysis 1: Comparison: Active Control-SAP vs KRX-0502 (Ferric Citrate)-SAP; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: IV Iron Analysis
Description: Full Analysis Population, cumulative IV Iron administration from Baseline to the end of the Safety Assessment Period (Week 52)
Time Frame: 52 weeks
Measure: Median (Full Range); unit: mg/day
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Number analyzed (Participants) | 138 | 271 | 0 | 0
mg/day | 3.83 [0.0 to 43.6] | 1.87 [0.0 to 24.2] |  |
Statistical Analysis 1: Comparison: Active Control-SAP vs KRX-0502 (Ferric Citrate)-SAP; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: ESA Analysis
Description: Full analysis population, cumulative Erythropoiesis-stimulating agent (ESA) administration from baseline to the end of the Safety Assessment Period (Week 52)
Time Frame: 52 weeks
Measure: Median (Full Range); unit: Units/Day
Arm/Group | Active Control-SAP | KRX-0502 (Ferric Citrate)-SAP | Placebo-EAP | KRX-0502 (Ferric Citrate)-EAP
Number analyzed (Participants) | 141 | 273 | 0 | 0
Units/Day | 993.46 [0.0 to 11015] | 755.80 [0.0 to 8171.9] |  |
Statistical Analysis 1: Comparison: Active Control-SAP vs KRX-0502 (Ferric Citrate)-SAP; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Serious treatement emergent adverse events (TEAEs) up to 56 weeks
Description: Safety Population, includes all patients that took at least 1 dose of study drug
Groups:
- KRX-0502 (SAP); Active Control (SAP): Safety Assessment Period (Week 1-52)
- KRX-0502 (EAP); Placebo (EAP): Efficacy Assessment Period (Week 52-56)
Arm/Group | KRX-0502 (SAP) | Active Control (SAP) | KRX-0502 (EAP) | Placebo (EAP)
Serious Adverse Events (participants affected / at risk) | 114/289 | 73/149 | 11/95 | 17/95
Other Adverse Events (participants affected / at risk) | 211/289 | 88/149 | 5/95 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRX-0502 (SAP) (N=289) | Active Control (SAP) (N=149) | KRX-0502 (EAP) (N=95) | Placebo (EAP) (N=95)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Graft thrombosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Blood and lymphatic system disorders) | 5 (5) | 8 (8) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Aortic stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Chest discomfort (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 8 (8) | 5 (5) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertensive crisis (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Sudden death (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Ileitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fluid Overload (General disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Hyperkalemia (General disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Hypokalemia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 | 0 (0)
Mental disorder (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Leg amputation (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal transplant (Surgical and medical procedures) | 13 (13) | 5 (5) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 5 (5) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 4 (4) | 1 (1) | 0 (0)
Vascular access complication (Vascular disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous Graft Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridial Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Graft Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diastolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrosis Ischaemic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Steal Syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adverse Event (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device Occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia Obstructive (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial Bypass Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous Fistula Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Debridement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreas Transplant (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal And Pancreas Transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stent Placement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural Hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain Stem Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheterisation Cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cancer Metastatic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Viral Infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Cyst Infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism And Nutrition Disorders (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary Disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy Hypertensive (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRX-0502 (SAP) (N=289) | Active Control (SAP) (N=149) | KRX-0502 (EAP) (N=95) | Placebo (EAP) (N=95)
Dyspnea (Cardiac disorders) | 10 (10) | 11 (11) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 14 (14) | 7 (7) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 21 (21) | 6 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 72 (72) | 19 (19) | 0 (0) | 0 (0)
Feces discolored (Gastrointestinal disorders) | 49 (49) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 38 (38) | 18 (18) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (24) | 18 (18) | 0 (0) | 0 (0)
Chest pain (General disorders) | 15 (15) | 6 (6) | 0 (0) | 0 (0)
Edema peripheral (General disorders) | 9 (9) | 8 (8) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 7 (7) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 21 (21) | 9 (9) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 12 (12) | 8 (8) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 23 (23) | 14 (14) | 5 (5) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 5 (5) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (8) | 9 (9) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (15) | 14 (14) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 14 (14) | 10 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 22 (22) | 11 (11) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 15 (15) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 7 (7) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 10 (10) | 0 (0) | 0 (0)
Hypotension (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 12 (12) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No